CLINICAL TRIAL: NCT06821594
Title: Role of Intralesional Combined Injection of Furosemide and Digoxin in Cutaneous Warts.
Brief Title: Role of Intralesional Combined Injection of Furosemide and Digoxin in Cutaneous Warts at Tertiary Care Hospital in Karachi.
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Rashida Kaizar, Postgraduate trainee, Jinnah Postgraduate Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2024-GENL/22/JPMC
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Warts
Keywords: Cutaneous warts; furosemide; digoxin
MeSH Terms: interventions — Furosemide; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients with age between 18-60 years having more than two cutaneous warts will be given combined intralesional furosemide (20mg/2ml) and digoxin (0.5mg/2ml) 0.2 ml at the base of warts once weekly for five weeks
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Furosemide 20mg/2ml and digoxin 0.5mg/2ml given 0.2 ml into the wart base once weekly for 5 weeks
  Other Names: Digoxin

SUMMARY:
Identify the effects of combined intralesional furosemide 20mg/2ml and digoxin 0.5mg/2ml in cutaneous warts given weekly are rather safe and effective treatment for cutaneous warts, focusing on their effectiveness and safety, at a tertiary care hospital in Karachi, Pakistan.

DETAILED DESCRIPTION:
Cutaneous warts are benign growth caused by human papilloma virus. Virus have more than 100 types of which few are responsible for cutaneous disease. Both injection furosemide and digoxin cause decrease intracellular potassium levels by interacting with cell membrane ion co-transporters (Na+/K+-ATPase and Na+-K+-2Cl-co-transporter-1) thereby causing delay in viral replication. The purpose of study is to evaluate the effects of both furosemide and digoxin given 0.2 ml once weekly for five weeks on viral warts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with greater than or equal to two warts
2. Either gender.
3. Age 18 - 60 years. -

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patient not giving informed consent.
3. Patient received any treatment in the last 3 months period.
4. Patient with acute illness and immuno-suppressive disease.
5. Patient taking immuno-suppressive drugs.
6. Patient having hypersensitivity to any investigational medicine.
7. Patient having cutaneous warts on face and genitals.
8. Patient having cardiovascular disease.
9. Patient having renal disease. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Size of cutaneous wart | 5 weeks
  Change in the dimensions of cutaneous wart assessed by Physician's wart assessment scale weekly and through photographs taking at the start and end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Intralesional combined digoxin and furosemide versus intralesional 5-flurouracil for the treatment of recalcitrant plantar warts: a prospective, randomized study — https://doi.org/10.1007/s00403-024-03014-z